CLINICAL TRIAL: NCT00282178
Title: A 36 Week Three-Center Double-Blind Randomized Cross-Over Trial Comparing Metabolic Effects of Candesartan, Hydrochlorothiazide and Placebo
Brief Title: Double-Blind Randomized Cross-Over Trial Comparing Metabolic Effects of Candesartan, Hydrochlorothiazide and Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Sahlgrenska University Hospital (Other); AstraZeneca (Industry)
Responsible Party: Jan Eriksson, Umeå University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2452L00007
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension; Obesity
Keywords: Metabolic; Hypertension; Abdominal obesity; Insulin sensitivity; Hyperinsulinemic euglycemic clamp
MeSH Terms: conditions — Hypertension; Obesity; Obesity, Abdominal; Insulin Resistance | interventions — Hydrochlorothiazide; candesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Candesartan 16-32 mg once daily
  Interventions: Drug: Candesartan
- 2 (Active Comparator): Hydrochlorothiazide 25-50 mg once daily
  Interventions: Drug: Hydrochlorothiazide
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrochlorothiazide — 25-50 mg once daily
  Arms: 2
Drug: Placebo — Once daily
  Arms: 3
Drug: Candesartan — 16-32 mg once daily 12 weeks
  Arms: 1

SUMMARY:
The purpose of this study is to investigate the effect of a 12-week candesartan treatment compared with hydrochlorothiazide on insulin sensitivity assessed with hyperinsulinemic euglycemic clamp.

DETAILED DESCRIPTION:
To investigate the mechanisms underlaying the diabetes-preventing effect of candesartan with respect to possible impact on insulin sensitivity, beta cell function and adipose tissue function and distribution. For this purpose comparisons will be performed with hydrochlorothiazide and placebo treatment. It is hypothesized that candesartan will improve insulin sensitivity as compared to hydrochlorothiazide and possibly also in comparison with placebo and that this could be explained by altered fat tissue function or distribution or by an altered sympathetic to parasympathetic balance in the autonomic nervous system. Hydrochlorthiazide is chosen as comparator because thiazides are a recommended firs-line therapy in hypertension. This drug class has some detrimental effects on glucose tolerance and in insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18-70 years old
* Diagnosed hypertension and abdominal obesity (waist circumference greater than or equal to 102 cm (M) or 88 cm (F)

Exclusion Criteria:

* Uncontrolled hypertension
* Treatment with more than two concomitant antihypertensive medications
* Diabetes Mellitus
* Other endocrine disorder
* Severe liver disease
* Severely reduced renal function
* Malignant disease
* Alcohol or drug abuse
* Severe psychiatric illness
* History of stroke, myocardial infarction, unstable angina pectoris, participation in another clinical trial less than two months prior to screening visit
* treatment with anti-obesity drugs
* anti-inflammatory drugs or immunosuppressive drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-04; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Compare the effect of candesartan and hydorclorothiszide treatment on insulin sensitivity assessed with hyperinsulinemic euglycemic clamp | 12 weeks

SECONDARY OUTCOMES:
Compare the effect of candesartan treatment with placebo on insulin sensitivity and compared with hydrochlorothiazide and placebo on: | 12 weeks
beta cell function | 12 weeks
vascular/endothelial function; | 12 weeks
lipolysis regulation | 12 weeks
autonomic nerve activity; | 12 weeks
abdominal fat tissue distribution; | 12 weeks
amount of lean body and fat mass; | 12 weeks
liver and muscle fat; | 12 weeks
interaction betw. insulin and AT-II in fat cell metabolism; fat cell gene expression | 12 weeks
adipokine levels | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eriksson, MD, PhD, Principal Investigator — Dept of Medicine, Umeå University Hospital, Sweden
Locations (1):
- Umeå University Hospital, Umeå, Sweden